CLINICAL TRIAL: NCT04090255
Title: Ultrasonography Versus Fluoroscopic Guided Renal Access
Brief Title: Us vs Fluoroscopic Guided Renal Access
Acronym: Puncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mostafa kamel abdel rahman abdel aal, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Renal puncture
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Hydronephrosis
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonographic guided renal access (Experimental): The use of ultrasound to make a puncture in kidney for pcn for drainage or evaluation of function or for shunt of urine
  Interventions: Procedure: Renal puncture
- Fluoroscopic guided renal access (Experimental): The use of fluoroscopy to make a puncture in kidney for pcn for drainage or evaluation of function or for shunt of urine
  Interventions: Procedure: Renal puncture

INTERVENTIONS:
Procedure: Renal puncture — The use of a needle for entering pelvicalyceal system of the kidney and put a guide wire for further pcn

SUMMARY:
this present study is to compare the result of fluoroscopy, ultrasonography (US) in the guidance of percutaneous nephrostomy pcn .

DETAILED DESCRIPTION:
investigators will enroll 100 patients who are candidates for PCN in the study. By simple random sampling technique, patients will be assigned to two patient groups (group 1, US-guided approach , group 2, fluoroscopy-guided approach.The end point of the study is the comparison of outcome of procedure including stone free rate, transfusion rate, operation time, access time, length of stay and complications.

ELIGIBILITY:
Inclusion Criteria:

* infected hydronephrotic kidney onen's grade 2-3
* obstructed good cortex with backpressure changes onen's grade 2-3 .
* Evaluation of function of asymptomatic hydronephrotic kidney thin cortex onen's grade 4

Exclusion Criteria:

* congenital anomalies of kidney
* patient underwent transplant or urinary diversion
* solitary kidney

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Duration of puncture | Within the operation
  The time taken for make a puncture
duration of operation | withen the operation
  time taken from patient putted on table until end of operation
Rate of success | withen the operation
  the rate success of intervention by u/s or by fluoroscopy

SECONDARY OUTCOMES:
rate of Perioperative complication | withen the operation
  numbers of patients with Adverse effects occures intra operative ,bleeding ,extravasation
Haemoglobin concentration change | 24 hours post procedure
  Compare preoperative and post operative Hg concentration

CONTACTS AND LOCATIONS:
Overall Officials: Fathy G Elanany, Prof, Study Director — Assiut; Mohamed A Sayed, Prof, Study Director — Assiut; Hosney M Bahnasawy, Ass Prof, Study Director — Assiut
Locations (1):
- Mostafs Kamel Abdel Rahman, Asyut, Sedfa, Egypt

REFERENCES:
- [Background] Chen X, Peng PX, He YH, Ding ZS, Wang JF, Tan YW, Zhou XF. [Evaluation and Comparison of SHA.LIN,S.T.O.N.E.Nephrolithometry Scoring System,and Clinical Research Office of the Endourological Society Nephrolithometry Nomogram for Predicting Stone Free Rate and Postoperative Outcomes after Percutaneous Nephrolithotomy]. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 2019 Aug 30;41(4):492-500. doi: 10.3881/j.issn.1000-503X.10767. Chinese. PMID 31484611
- [Background] Zanetti SP, Boeri L, Gallioli A, Talso M, Montanari E. Minimally invasive PCNL-MIP. Arch Esp Urol. 2017 Jan;70(1):226-234. PMID 28221157
- [Background] Gulati M, Cheng J, Loo JT, Skalski M, Malhi H, Duddalwar V. Pictorial review: Renal ultrasound. Clin Imaging. 2018 Sep-Oct;51:133-154. doi: 10.1016/j.clinimag.2018.02.012. Epub 2018 Feb 16. PMID 29477809
- [Background] Qiu Z, Yang Y, Zhang Y, Sun YC. Modified biological training model for percutaneous renal surgery with ultrasound and fluroscopy guidance. Chin Med J (Engl). 2011 May;124(9):1286-9. PMID 21740734